CLINICAL TRIAL: NCT06434558
Title: Imaging Predictors of Cryolysis Efficacy for Treatment of Obstructive Sleep Apnea
Acronym: ICE-OSA
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Raj Dedhia, MD, Associate Professor of Otorhinolaryngology & Medicine | Director, Division of Sleep Surgery & CPAP Alternatives Clinic, University of Pennsylvania
Other Study IDs: 855200
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: Obstructive Sleep Apnea; ultrasound; MRI; cryotherapy
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Cryotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cryosa Procedure — The Cryosa Procedure is part of the ARCTIC-3 protocol (IRB #854182). Therefore, all patients enrolled in this study are expected to undergo the Cryosa Procedure. Undergoing the Cryosa Procedure is not a part of this protocol.
  Other Names: Cryotherapy; OSA Cryotreatment

SUMMARY:
The goal of this observational study is to further evaluate the efficacy and mechanism of action of the Cryosa Procedure, a novel procedure intended to treat obstructive sleep apnea (OSA). The patient population includes participants with OSA who are enrolled in the ARCTIC-3 study and are undergoing the Cryosa Procedure. The main questions to be answered are:

(1) evaluate predictors of successful treatment with the Cryosa Procedure, which is described in more detail in the ARCTIC-3 protocol (IRB #854182), and (2) evaluate a potential mechanism of action of this novel therapy.

The study team hypothesizes that higher baseline quantities of oropharyngeal fat and higher baseline upper airway neurotonic activity will be correlated with a successful reduction in OSA symptom severity as measured by a change in apnea-hypopnea index values. The study team also hypothesizes that responders will have a decrease in oropharyngeal fat, which would indicate the mechanism of action of this novel therapy is a loss in oropharyngeal fat.

Participants will be asked to:

1. have an MRI before undergoing the Cryosa Procedure
2. have an ultrasound before the Cryosa Procedure
3. permit the use of pressure-sensing catheters and ultrasound during their drug-induced sleep endoscopy, which is part of the ARCTIC-3 protocol
4. have an MRI after the Cryosa Procedure
5. have an ultrasound after the Cryosa Procedure.

DETAILED DESCRIPTION:
Previous research has shown there is increased fat at the base of the tongue and other locations of the oropharynx in patients with Obstructive Sleep Apnea (OSA) compared to match control non-OSA patients. Subsequently, Cryosa developed the Cryosa Procedure, which is further detailed in the ARCTIC-3 protocol (IRB #854182). This procedure involves the Cryosa System, a device intended to induce adipose cryolysis, a non-surgical removal of by inducing cell death (apoptosis) with a controlled freezing of the soft tissue, in the upper airway.

Whereas the objective of the ARCTIC-3 study is to determine the efficacy and safety of the Cryosa Procedure, the co-primary aims of the ICE-OSA study are to (1) evaluate predictors of successful treatment with the Cryosa Procedure and (2) evaluate a potential mechanism of action of this novel therapy. The study team hypothesizes that (1) higher baseline quantity of oropharyngeal fat and higher baseline upper airway neurotonic activity are correlated with a successful reduction in OSA severity, and (2) responders will have a decrease in quantity of oropharyngeal fat (as measured by post-operation magnetic resonance imaging, MRI). Investigating the mechanisms and predictors of this novel therapy is necessary to inform future clinical trials and patient selection for the Cryosa Procedure. To assess these metrics, the ICE-OSA study utilizes MRI, point-of-care ultrasound (POCUS), and the addition of pharyngeal manometry and ultrasound (US) during drug-induced sleep endoscopy (DISE) for ARCTIC-3 participants.

Study Statistics:

These prognostic data are going to be collected as part of a small pilot study to inform the upcoming pivotal trial. For this reason, investigators seek independent variables with large effect sizes to update and enhance patient selection criteria for the future trial.

The study team propose use of Student's t-test for responders/non-responders (responder defined as reduction of AHI by >50%) for the surgical intervention. The expected ratio of responders to non-responders is 1:1 based on data provided by the study sponsor (unpublished).

Previous data examining tongue fat in MRI demonstrated values of quantity of fat tissue in fatty tongues to be roughly 14,000 mm3 and fat tissue in non-fatty tongues to be roughly 7,000 mm3. Using these parameters, it was calculated that 10 subjects total would be required (assuming a standard deviation of 4,000 mm3) to detect significant differences between responders/non-responders with an alpha of 0.05 and a power of 80%.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the ARCTIC-3 clinical trial at the University of Pennsylvania*
* Provision of signed and dated informed consent form for ICE-OSA

Exclusion Criteria:

* MRI contraindications (claustrophobia, ferromagnetic implants/foreign bodies, etc.)
* Patient is pregnant or becomes pregnant during their enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study enrolls only participants that are previously enrolled in the ARCTIC-3 trial and are subsequently undergoing the Cryosa Procedure as part of the ARCTIC-3 protocol. As required by the eligibility criteria in the ARCTIC-3 study, these patients have a BMI less than or equal to 40 kg/m2, are 22 to 70 years old, and have moderate to severe obstructive sleep apnea (OSA).
  Additionally, eligibility requirements from the ARCTIC-3 trial include having never previously undergone uvulopalatopharyngoplasty or tongue base reduction for the treatment of OSA. Patients are also excluded for any other reasons the principal investigator would deem a contraindication to undergoing procedures outlined by the ARCTIC-3 protocol.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Oropharyngeal Fat at 6 Months | Baseline and 6 months
  Quantity of oropharyngeal fat will be measured with magnetic resonance imaging (MRI) before the Cryosa Procedure and 6 months after the Cryosa Procedure in all subject participants.
Change in Baseline Apnea Hypopnea Index at 6 Months | Baseline and 6 Months
  All participants in this study, who are also enrolled in the ARCTIC-3 study, are undergoing a polysomnogram as part of the ARCTIC-3 study at baseline and at 6 months. AHI is measured during these sleep studies in every patient at both timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Raj Dedhia, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT06434558/ICF_000.pdf